CLINICAL TRIAL: NCT07042711
Title: Effect of Vitamin D Supplementation on Therapeutic Response in Nasopharyngeal Cancer (NPC) Patients Undergoing Chemoradiation and Its Relation With IL-6
Brief Title: Impact of Vitamin D on Therapeutic Respons in NPC Chemoradiated Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Budi Wiweko, Clinical Professor, Indonesia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS01
Record Dates: First submitted 2025-06-12; First posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Nasopharyngeal Cancinoma (NPC)
Keywords: Vitamin D; Nasopharyngeal Cancer; NPC; Human Interleukin-6; Chemoradiation; Therapy; HIL-6; Radioteraphy
MeSH Terms: conditions — Nasopharyngeal Neoplasms | interventions — Vitamin D; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vitamin D Group (Experimental): NPC patients received capsules containing vitamin D or a placebo to the and neither patient nor researcher knows
  Interventions: Dietary Supplement: Placebo; Dietary Supplement: Vitamin D 5,000IU Oral Tablet

INTERVENTIONS:
Dietary Supplement: Placebo — Patients are given capsules that can contain either a placebo or Vitamin D.
  Other Names: Control
Dietary Supplement: Vitamin D 5,000IU Oral Tablet — Patients are given capsules that can contain either a placebo or Vitamin D.

SUMMARY:
Nasopharyngeal cancer is the sixth most common cancer and the sixth leading cause of death in Indonesia. NPC is a radiosensitive cancer so radiotherapy is the basic therapy for NPC. Concurrent chemoradiotherapy (CCRT) with Intensity modulated radiotherapy (IMRT) is the standard therapy for locally advanced NPC. Vitamin D deficiency is common in patients with head and neck cancer including NPC. Several studies have shown better outcomes and fewer complications of therapy in patients with higher vitamin D levels. Inflammation plays an important role in tumor development and progression. The effect of vitamin D supplementation on cancerous and precancerous lesions shows that there is a potential for major changes in IL-6 levels.

By supplementing vitamin D in NPC patients with vitamin D deficiency before undergoing chemoradiation, it will increase the therapeutic response and reduce IL-6 levels (proinflammatory cytokines). Until now, there have been no studies evaluating the administration of vitamin D supplementation in NPC patients with vitamin D deficiency undergoing chemoradiation in Indonesia.

DETAILED DESCRIPTION:
According to the Global Cancer Observatory (Globocan) 2022, nasopharyngeal cancer (NPC) is the sixth most common cancer and the sixth leading cause of death among all cancers in Indonesia. The incidence of NPC varies across regions of the world, with the highest incidence for men and women detected in Southeast Asia (7.7 and 2.5 per 100,000 person-years, respectively), in Indonesia itself the NPC incidence rate is 10.7 per 100,000 person-years and the mortality rate is 7.7 per 100,000 person-years. NPC is a radiosensitive cancer so radiotherapy is the basic therapy for NPC. The outcome of NPC patient treatment has improved over the past decade, especially after the introduction of Concurrent chemoradiotherapy (CCRT) with Intensity modulated radiotherapy (IMRT) and induction chemotherapy. Patients who receive radiotherapy with IMRT will provide better therapeutic results with milder long-term side effects than conventional radiotherapy techniques. Vitamin D deficiency is more common in head and neck cancer patients compared to healthy populations. Vitamin D can downregulate the expression of nuclear factor kappa light chain enhancer of activated B cells (NF-κB) and also inhibit the inflammatory response mediated by immune cells through the vitamin D receptor (VDR) expressed on human cells. Several studies have shown the tumor suppressive effect of vitamin D through antitumor activity in various cancers. Vitamin D also has a role in potentiating antitumor activity through radiotherapy. IL-6 is a pro-inflammatory cytokine that plays an important role in the TME. Serum IL-6 levels in NPC patients increase and correlate with advanced stages. Low vitamin D levels before therapy are associated with worse outcomes and increased treatment-related complications, so it is important to manage vitamin D deficiency in NPC patients to improve the response to therapy.

ELIGIBILITY:
Inclusion Criteria:

* NPC stage III-IVA who will undergo chemoradiation
* Have vitamin D deficiency (vitamin D level <30 ng/mL)
* Age > 18 years
* WHO ECOG performance status 0-2

Exclusion Criteria:

* Subject has autoimmune disease
* Subject is undergoing immunosuppressive therapy
* Patient routinely consumes vitamin D supplementation
* Experiencing other acute conditions (eg: severe infection)
* Subject cannot be evaluated (drop out, loss to follow up)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2025-12-09 (Estimated); Study Completion 2025-12-09 (Estimated)

PRIMARY OUTCOMES:
Effect of Vitamin D Supplementation on therapeutic response in nasopharyngeal cancer (NPC) patients undergoing chemoradiation and its relation with IL-6 | January 2025 - Juny 2025
  Therapeutic response is evaluated using RECIST 1.1 criteria based on MRI findings, and categorized into favorable response (Complete Response [CR] and Partial Response [PR]) and poor response (Stable Disease [SD] and Progressive Disease [PD]). The main outcome is the difference in response between groups

SECONDARY OUTCOMES:
Effect of Vitamin D Supplementation on therapeutic response in nasopharyngeal cancer (NPC) patients undergoing chemoradiation and its relation with IL-6 | January 2025 - Juny 2025
  To compare the mean change in serum IL-6 levels (pg/mL) from Pre-chemoradiation to post-chemoradiation between participants receiving placebo and those receiving vitamin D supplementation.

CONTACTS AND LOCATIONS:
Overall Officials: Budi Wiweko, MD, Principal Investigator — Indonesia University
Locations (1):
- Dr Cipto Mangunkusumo Hospital and Dharmais Cancer Hospital, Jakarta, Jakarta Special Capital Region, Indonesia

IPD SHARING:
Plan to Share IPD: No